CLINICAL TRIAL: NCT04239690
Title: A Randomised Controlled Intervention, Multi-centre Study Aiming to Preserve Blood Factors Using Micro-methods to Improve Development in Extremely Preterm Infants - "Less is More"
Brief Title: Preservation of Blood in Extremely Preterm Infants
Acronym: LIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Ley (Other)
Responsible Party: Sponsor-Investigator, David Ley, Professor, Lund University
Organization: Lund University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018-00770
Record Dates: First submitted 2020-01-19; First posted 2020-01-27 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Extremely preterm infant; Blood sampling; Blood transfusion
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Outcomes Assessor
Masking Description: Prevalence and severity of BPD at 36 weeks post-menstrual age is determined by the oxygen challenge test performed by a trained respiratory nurse blinded to treatment at each study site.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Micromethods for blood sample analysis (Experimental): Blood gases are analysed using 0.045 ml whole blood Levels of C-reactive protein (CRP) are analysed using 0.010 ml whole blood
  Interventions: Other: Micromethods for blood sample analysis
- Standard clinical methods for blood sample analysis (No Intervention): Blood gases are analysed using 0.3 ml whole blood Levels of CRP are analysed using 0.5 ml whole blood

INTERVENTIONS:
Other: Micromethods for blood sample analysis — Micromethods in the intervention arm are applied aiming to achieve a mean reduction of 50 % of sampled blood volume during the first two postnatal weeks as compared to standard clinical blood sampling analyses
  Arms: Micromethods for blood sample analysis

SUMMARY:
Current clinical protocols for blood sampling and analyses in extremely preterm infants rely on an infrastructure adapted to and developed for adult medicine. Excessive blood sampling volumes and the resulting loss of fetal blood components are related to neonatal morbidity. This randomised trial aims to provide evidence that preservation of blood using micro-methods results in decreased morbidity and increased quality of life in extremely preterm infants.

DETAILED DESCRIPTION:
Extremely preterm (EPT) infants are subjected to a sample-related withdrawal of whole blood of 50 % of total blood volume during the first 2 postnatal weeks and a transfused volume of 100 % of total blood volume with donor blood during the corresponding time period. The resulting decrease in the proportion of fetal hemoglobin is strongly associated with morbidity outcome, especially broncho-pulmonary dysplasia (BPD), in the EPT infant.

This randomized trial evaluates if a reduction in sample-related blood volume loss by 50% during the first two postnatal weeks leads to a reduced rate of BPD in EPT infants. Half of the included infants will be subjected to clinical blood sampling using micromethods during the first two postnatal weeks whereas blood sampling in the other half of infants will be performed using standard clinical methods.

ELIGIBILITY:
Inclusion Criteria:

* gestational age < 27 weeks at birth

Exclusion Criteria:

* major malformation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Broncho-pulmonary dysplasia | Broncho-pulmonary dysplasia is determined at a postmenstrual age of 36 weeks
  Requirement of supplemental oxygen as determined by the oxygen challenge test

SECONDARY OUTCOMES:
Cerebral intraventricular haemorrhage | Ultrasound at postnatal day 3, 7, 21 and 40 weeks postmenstrual age
  Stage II, III and IV (Periventricular hemorrhagic infarction)
Necrotizing enterocolitis | From birth until 40 weeks postmenstrual age
  Stage 2-3, Bells criteria (X-ray + clinical signs)
Blood transfusions | Blood transfusions administered during the first two postnatal weeks
  Administered blood transfusions (ml/kg)
Fetal Hemoglobin | % of fetal hemoglobin at 7 and 14 postnatal days
  % of fetal hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: David Ley, MD, PhD, Principal Investigator — Lund University, Lund, Sweden
Locations (1):
- Neonatal Intensive Care Unit, Lund, Sweden

REFERENCES:
- [Derived] Larsson SM, Ulinder T, Rakow A, Vanpee M, Wackernagel D, Savman K, Hansen-Pupp I, Hellstrom A, Ley D, Andersson O. Hyper high haemoglobin content in red blood cells and erythropoietic transitions postnatally in infants of 22 to 26 weeks' gestation: a prospective cohort study. Arch Dis Child Fetal Neonatal Ed. 2023 Nov;108(6):612-616. doi: 10.1136/archdischild-2022-325248. Epub 2023 May 11. PMID 37169579
- [Derived] Hellstrom W, Martinsson T, Morsing E, Granse L, Ley D, Hellstrom A. Low fraction of fetal haemoglobin is associated with retinopathy of prematurity in the very preterm infant. Br J Ophthalmol. 2022 Jul;106(7):970-974. doi: 10.1136/bjophthalmol-2020-318293. Epub 2021 Feb 5. PMID 33547036